CLINICAL TRIAL: NCT02145169
Title: Inhaled Nitrous Oxide for the Prevention of Emergence Reaction During Ketamine Administration in Adults, a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HN4507FBD
Record Dates: First submitted 2014-05-09; First posted 2014-05-22 (Estimated); Results first posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2016-12

CONDITIONS: Emergence Reaction; Procedural Sedation
Keywords: procedural sedation; emergence reaction; nitrous oxide; ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nitrous Oxide arm (Experimental): Patients will receive a 50/50 mixture of Oxygen and Nitrous oxide via non breather mask
  Interventions: Drug: Inhaled Nitrous Oxide

INTERVENTIONS:
Drug: Inhaled Nitrous Oxide — Patients undergoing procedural sedation with Ketamine will receive inhaled Nitrous Oxide

SUMMARY:
To describe the safety and efficacy of nitrous oxide during ketamine administration for the prevention of emergence reaction during Emergency Department procedural sedation and analgesia in adults. Drugs such as fentanyl, midazolam, and propofol are widely used in emergency departments for procedural sedation and analgesia because they have a rapid onset and short duration of action. Unfortunately, all of these agents may cause respiratory depression, particularly when combined with other sedative agents, administered in large doses, or given to patients with underlying respiratory diseases. Nitrous oxide use during ketamine administration may be an ideal combination for the prevention of emergence reaction in adults sedated in the ED. Like ketamine, nitrous oxide has an excellent cardio-respiratory profile as well as some analgesic and anxiolytic qualities. The anxiety and pain surrounding procedural sedation is not limited to the procedure itself, but the elapsed time from the time the patient enters the ED to the time spent in preparation for the procedure can be significant and lead to increased anxiety, which may exacerbate emergence reactions in adults. Using nitrous oxide before ketamine administration may mitigate this. While midazolam has shown efficacy in reducing emergence reactions in adults sedated with ketamine, the investigators believe that inhaled nitrous oxide may be equivalent to midazolam, with a better cardio-respiratory profile.

DETAILED DESCRIPTION:
Drugs such as fentanyl, midazolam, and propofol are widely used in emergency departments for procedural sedation and analgesia because they have a rapid onset and short duration of action. Unfortunately, all of these agents may cause respiratory depression, particularly when combined with other sedative agents, administered in large doses, or given to patients with underlying respiratory diseases.

Ketamine hydrochloride is a phencyclidine derivative that causes dissociation between the cortical and limbic systems preventing the higher centers from perceiving visual, auditory, or painful stimuli. It possesses a rapid onset and short duration of action and produces profound sedation and analgesia. Ketamine is also a non-competitive NMDA antagonist, which complements NO. However, laryngeal reflexes are maintained and respiratory depression is rare. These properties have made ketamine a very popular agent for procedural sedation and analgesia in pediatric emergency department patients . Unfortunately, when given to adult patients, it frequently causes emergence anxiety, nightmares, hallucinations, and delirium. These emergence reactions have limited the use of ketamine in adults. The incidence of these reactions is about 7-10% in children. Emergence reactions may be a product of the state in which the patient becomes disassociated . Therefore, if the patient is more relaxed prior to ketamine administration through the adjunct use of NO, adverse emergence reactions may be reduced.

A number of agents including diazepam, lorazepam, fentanyl, droperidol, and others have been used with varying success to reduce or prevent emergence reactions associated with ketamine use. Diazepam and lorazepam have been the most successful, but their use may prolong recovery time, making them less desirable in the emergency department setting. Midazolam has been shown to lower the rate of emergence reaction when used concurrently with ketamine in adults. However, like all benzodiazepines, there is a small risk of respiratory depression and hypoxia with the use of midazolam, which could lead to an adverse respiratory event.

Inhaled nitrous oxide may be an ideal adjunct to the prevention of emergence reaction in adults being treated with ketamine. Nitrous oxide is a colorless gas that diffuses rapidly across the pulmonary alveoli providing analgesia and anxiolysis with minimal sedative effects, rapid induction, and emergence. Nitrous oxide is a weak sedative agent with the potential for significant analgesic effects. Noncompetitive antagonist activity at the NMDA receptor along with activation of opioid receptors contributes to its anesthetic mechanism. There are rare adverse events, most often cited as case reports of chronic or acute toxicity causing myeloneuropathies and polyneuropathies.

Nitrous oxide has been used in general anesthesia for over 2 centuries, but its use outside of the operating room began when Tunstall introduced the nitrous oxide/oxygen mixture as an analgesic agent during labor. Since this inception, the nitrous oxide/oxygen mixture has been used readily in the fields of dentistry, gastrointestinal procedures, and children's procedural sedation. Nitrous oxide is often administrated via continuous flow or on-demand at a concentration of 50-70%.

There is some early data describing a favorable adverse event profile with nitrous oxide as a single agent in adults. Hennequin et al. demonstrated support for the efficacy of nitrous oxide with no major adverse cardio respiratory events. Although approximately 10% of participants received mild gastrointestinal and behavioral side effects (e.g. agitation). Greater than 90% of the study participants stated they would receive nitrous oxide again. In a large prospective trial, Babl et al. found there to be only 2 patients out of 655 who suffered serious adverse events (i.e., chest pain and oxygen desaturation). Both patients had been administered 70% nitrous oxide compared to the more conservative 50% concentration. Additionally, there was an increased incidence of minor adverse events (i.e., emesis and agitation) with the higher concentration of nitrous oxide. Kariman et al. compared nitrous oxide versus parental fentanyl as an analgesic after long bone fracture and found similar pain scores and a more rapid decrease in the pain score in the nitrous oxide group when compared with the opiate group.

Nitrous oxide has been shown to be a safe and effective agent for procedural sedation in children, including work that has combined opiates and benzodiazepines with nitrous continuously. Burton et al. conducted a small, randomized controlled trial studying the effectiveness of nitrous oxide on anxiety scores in children during laceration repairs. They found a significant decrease in the group that used nitrous oxide compared to the placebo group. This finding was further validated by Luhmann et al. with 50% continuous flow nitrous oxide resulting in less distress and anxiety as well as increased patient satisfaction compared to midazolam or topical anesthetic agents. The study also showed that the main adverse event associated with nitrous oxide was nausea and vomiting, whereas midazolam group had significant ataxia and dizziness. There was no demonstrable advantage of the combination of midazolam and nitrous oxide in regard to patient satisfaction versus nitrous oxide alone, but there was an increase in adverse events when midazolam was included.

A study performed by Evans et al. demonstrated that the pain and memory of the procedure between children receiving either nitrous oxide versus children receiving intramuscular meperidine in combination with promethazine for fracture reduction was similar, but there was increased satisfaction and decreased length of stay in the nitrous oxide group. Seith et al. demonstrated that the addition of intranasal fentanyl to nitrous oxide in children resulted in deeper levels of sedation when compared to nitrous oxide alone; however, there were no serious adverse events.

Nitrous oxide use during ketamine administration may be an ideal combination for the prevention of emergence reaction in adults sedated in the ED. Like ketamine, nitrous oxide has an excellent cardio-respiratory profile as well as some analgesic and anxiolytic qualities. The anxiety and pain surrounding procedural sedation is not limited to the procedure itself, but the elapsed time from the time the patient enters the ED to the time spent in preparation for the procedure can be significant and lead to increased anxiety, which may exacerbate emergence reactions in adults. Using nitrous oxide before ketamine administration may mitigate this. While midazolam has shown efficacy in reducing emergence reactions in adults sedated with ketamine, we believe that inhaled nitrous oxide may be equivalent to midazolam, with a better cardio-respiratory profile.

Since this is a novel concept, we believe that a pilot study to evaluate the safety and efficacy of 50/50 nitrous oxide/oxygen administration with adult ketamine administration is warranted.

ELIGIBILITY:
Inclusion criteria: All spontaneously breathing subjects, 18 years of age and older, with an American Society of Anesthesiologists (ASA) Physical Status Classification 1 or 2, who will be receiving sedation for an ED procedure. Written informed consent will be obtained from all subjects.

Exclusion criteria: Subjects with underlying conditions that could affect ventilation, perfusion, or metabolism including intubated subjects, subjects with clinical signs of cardiopulmonary instability, major trauma, thoracic trauma, shock, sepsis, psychiatric disorders and ASA class 3, 4, and 5. Also those unable to provide informed consent, nursing home residents, age less than 18 years, non English speaking, pregnant women, subjects under police custody, or physician discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Dominici, MD, Principal Investigator — Albert Einstein Healthcare Network
Locations (1):
- Albert Einstein Healthcare Network, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Pre-assignment Details: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Period: Overall Study
Arm/Group | Nitrous Oxide Arm
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Nitrous Oxide Arm
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Emergence Reaction
Description: Presence or absence of emergence reaction
Time Frame: At primary ED visit when the patient is undergoing the intervention
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Nitrous Oxide Arm
Number analyzed (Participants) | 0

2. Secondary Outcome: Physiologic Measure
Description: ETCO2 measured q 5 seconds
Time Frame: At primary ED visit when the patient is undergoing the intervention
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Nitrous Oxide Arm
Number analyzed (Participants) | 0

3. Secondary Outcome: Physiologic Measure
Description: SpO2 measured q 5 seconds
Time Frame: At primary ED visit when the patient is undergoing the intervention
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Nitrous Oxide Arm
Number analyzed (Participants) | 0

4. Secondary Outcome: Vitals
Description: heart rate, respiratory rate, peripheral SaO2
Time Frame: At primary ED visit when the patient is undergoing the intervention
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Nitrous Oxide Arm
Number analyzed (Participants) | 0

5. Secondary Outcome: Physician Interventions
Description: verbal or physical stimulation, airway repositioning, additional oxygen, positive pressure ventilation, endotracheal intubation
Time Frame: At primary ED visit when the patient is undergoing the intervention
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Nitrous Oxide Arm
Number analyzed (Participants) | 0

6. Secondary Outcome: Level of Sedation
Description: Ramsay sedation score
Time Frame: At primary ED visit when the patient is undergoing the intervention
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Nitrous Oxide Arm
Number analyzed (Participants) | 0

7. Secondary Outcome: Patient Recall of Procedure
Description: Patient recall of procedure
Time Frame: At primary ED visit when the patient is undergoing the intervention
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Nitrous Oxide Arm
Number analyzed (Participants) | 0

8. Secondary Outcome: Total Ketamine Dose
Description: Total Ketamine dose
Time Frame: At primary ED visit when the patient is undergoing the intervention
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Nitrous Oxide Arm
Number analyzed (Participants) | 0

9. Secondary Outcome: Total Time of Nitrous Use
Description: Total elapsed time of nitrous use
Time Frame: At primary ED visit when the patient is undergoing the intervention
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Nitrous Oxide Arm
Number analyzed (Participants) | 0

10. Secondary Outcome: Physician Procedure Satisfaction Score
Description: Physician procedure satisfaction survey responses
Time Frame: At procedure completion
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Nitrous Oxide Arm
Number analyzed (Participants) | 0

11. Secondary Outcome: Patient Procedure Satisfaction Score
Description: Patient procedure satisfaction survey responses
Time Frame: At procedure completion
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Nitrous Oxide Arm
Number analyzed (Participants) | 0

12. Secondary Outcome: Nurse Procedure Satisfaction Score
Description: Nurse procedure satisfaction survey responses
Time Frame: At procedure completion
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Nitrous Oxide Arm
Number analyzed (Participants) | 0

13. Secondary Outcome: Length of ED Stay
Description: Length of ED stay
Time Frame: At primary ED visit
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Nitrous Oxide Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 0
Description: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Nitrous Oxide Arm
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes